CLINICAL TRIAL: NCT02850133
Title: Effect of Aerobic Exercise Training on the Blood Biochemical Factors and Peripheral Hemodynamics in Person With Spinal Cord Injury
Brief Title: Aerobic Exercise and Blood Biochemical Factors in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201007031R
Record Dates: First submitted 2016-07-01; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal cord injury (Experimental): Cardio-pulmonary exercise testing and aerobic exercise training
  Interventions: Other: aerobic exercise training

INTERVENTIONS:
Other: aerobic exercise training — aerobic exercise training for 36 sessions within 12-16 weeks

SUMMARY:
Background:

Patients with spinal cord injury (SCI) have a higher prevalence of cardiovascular diseases compared to the healthy population. Aerobic exercise training is one of the recommended treatments. However, literature regarding the effect of aerobic training on patients with SCI is scarce. This study evaluated changes in parameters of exercise physiology and serum myokines immediately after exercise and after a training program among patients with SCI.

Method:

Male patients with SCI and age- and sex-matched healthy individuals were recruited. Cardio-pulmonary exercise testing (CPET) was used to determine oxygen uptake at peak exercise and anaerobic threshold in both groups. The patients with SCI attended aerobic exercise training for 36 sessions within 12-16 weeks. Basic data, hemodynamic and exercise physiology parameters, and serum myokine (myostatin, insulin like growth factor, and follistatin) concentrations were measured pre- and post-exercise in both groups, and were repeated in patients with SCI post-training.

DETAILED DESCRIPTION:
The patients with SCI were invited to undergo a 12- to 16-week exercise training by arm ergometry. The exercise physiology and measurements of hemodynamic parameters and cytokines were repeated after completion of the training.

ELIGIBILITY:
Inclusion Criteria:

* age >20 years, male sex, and onset of injury more than one year

Exclusion Criteria:

* known heart disease, atrial fibrillation/flutter, ventricular bigeminy, active inflammatory disease, malignancy, and cardiac pacemakers

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
serum myokines | 12-16 weeks

IPD SHARING:
Plan to Share IPD: Yes
The study is registered in publicly accessible site.